CLINICAL TRIAL: NCT04778033
Title: The Effect of BNT162b2 mRNA COVID-19 Vaccine on Semen Analysis Parameters Among 75 Fertile Men
Brief Title: Semen Analysis Parameters Following Pfizer's COVID-19 Vaccine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Jigal Haas MD, Senior Gynecologist and Obstetrician, Sheba Medical Center
Other Study IDs: SHEBA - 21 - 8079- JH - CTIL
Record Dates: First submitted 2021-02-08; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Fertility Issues
MeSH Terms: conditions — COVID-19; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Semen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccinated Men: Fertile men who were vaccinated with the BNT162b2 COVID-19 Vaccine
  Interventions: Other: Sperm collection

INTERVENTIONS:
Other: Sperm collection — Those recruited will supply a single sperm sample 1-2 months following the second dose of the vaccination. The sample will be analyzed for macroscopic and microscopic features in the IVF laboratory and will be discarded immediately afterwards.

SUMMARY:
In this study the investigators will explore the effect of the BNT162b2 COVID-19 Vaccine on semen analysis parameters among 75 fertile men. Fertile men will be regarded as such if they previously successfully impregnated their partners without the use of artificial reproductive technology, or men who previously had a normal sperm analysis exam by WHO criteria (2010). Those recruited will supply a single sperm sample 1-2 months following the second dose of the vaccination. In addition, the participants will fill a brief questionnaire with information regarding their medical and reproductive history. The investigators will examine the macroscopic and microscopic properties of the semen samples and compare them to the WHO semen analysis reference range in an attempt to ascertain whether the vaccine influences sperm parameters.

DETAILED DESCRIPTION:
The 2019 novel coronavirus disease (COVID-19) is a highly infectious respiratory tract disease which was first reported in Wuhan, Hubei Province, China in Dec 2019, but has since spread globally. By march 2020 it was declared by WHO as a public health emergency pandemic and has thus far affected tens of millions worldwide. The implications of COVID 19 infection on male fertility were examined in a previous study, which found decreased sperm concentration in recovering patients compared with controls.

The newly available mRNA COVID 19 vaccine by Pfizer was recently evaluated in a large multicenter placebo controlled RCT. The vaccine is comprised of BNT162b2, a lipid nanoparticle formulated nucleoside-modified RNA (modRNA) encoding the SARS-CoV2 full length spike protein, modified by two Proline mutations. The two 20 µg doses were shown to elicit high SARS-COV2 neutralizing antibody titers alongside high antigen specific CD8+ and Th1 type CD4+ T cell response. It was subsequently shown to be 95% effective in preventing COVID-19 infection a week following the second dose with a favorable safety profile in a 2-month median following up time.

Unfounded claims in the popular media linked a possible correlation between the COVID-19 vaccine and potential female\male infertility. Currently. there is no information in the medical literature which examined semen analysis parameters following the COVD-19 vaccine.

In this study the investigators will explore the effect of the BNT162b2 COVID-19 Vaccine on semen analysis parameters among 75 fertile men. Fertile men will be regarded as such if they previously successfully impregnated their partners without the use of artificial reproductive technology, or men who previously had a normal sperm analysis exam by WHO criteria (2010). Those recruited will supply a single sperm sample 1-2 months following the second dose of the vaccination. In addition, the participants will fill a brief questionnaire with information regarding their medical and reproductive history. The investigators will examine the macroscopic and microscopic properties of the semen samples and compare them to the WHO semen analysis reference range in an attempt to ascertain whether the vaccine influences sperm parameters.

ELIGIBILITY:
Inclusion Criteria:

* Previously impregnated their partner without the use of assisted reproduce technology, or previously had a normal sperm analysis exam by WHO 2010 criteria.
* 1-2 months following the second dose of BNT162b2 COVID-19 Vaccine.

Exclusion Criteria:

* Known abnormal semen parameters.
* Age above 45.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fertile men 1-2 months following the second dose of BNT162b2 COVID-19 Vaccine
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-04-10 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Sperm Concentration (10^6/ml) | 1-2 months after the second COVID-19 vaccine
  Semen concentration (10^6/ml)
Sperm Motility (%) | 1-2 months after the second COVID-19 vaccine
  Sperm percentage with proper forward progression
White Blood Cells (10^6/ml) in Semen | 1-2 months after the second COVID-19 vaccine
  Amount of white blood cells (10^6/ml) in semen
Sperm Morphology (%) | 1-2 months after the second COVID-19 vaccine
  Sperm morphology (%)
Sperm Vitality (%) | 1-2 months after the second COVID-19 vaccine
  Sperm vitality (%)
Semen Liquefaction (normal/abnormal) | 1-2 months after the second COVID-19 vaccine
  Macroscopic appearance - Semen liquefaction appearance
Semen Viscosity (normal/abnormal) | 1-2 months after the second COVID-19 vaccine
  Macroscopic appearance - Semen viscosity appearance
Semen Color | 1-2 months after the second COVID-19 vaccine
  Macroscopic appearance - Semen color appearance
Semen PH | 1-2 months after the second COVID-19 vaccine
  Semen PH
Semen Volume (ml) | 1-2 months after the second COVID-19 vaccine
  Semen Volume (ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No